CLINICAL TRIAL: NCT06761547
Title: Comparsion of Intravenous Injection of Magnesium Sulfate and Lidocaine Effectiveness on the Prevention of Laryngospasm and Analgesic Requirement in Tonsillectomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Monwar Shawky, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tonsillectomy operation
Record Dates: First submitted 2025-01-06; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (Active Comparator): patients will take magnsium sulfate 15 mg/kg on 50 ml saline
  Interventions: Drug: magnsium sulfate; Drug: Saline
- Group B (Active Comparator): Patients will take lidocaine2% 1 mg/kg on 50 ml saline
  Interventions: Drug: Lidocaine (drug); Drug: Saline
- Group c (Placebo Comparator): patients will take 50 ml saline only
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: magnsium sulfate — patients will take magnsium sulfate 15 mg/kg IV
  Arms: Group A
Drug: Lidocaine (drug) — patients will take lidocaine2% 1 mg/kg
  Arms: Group B
Drug: Saline — 50 ml saline IV

SUMMARY:
Tonsillectomy is one of the most common surgeries in children which is associated with many morbidities such as postoperative pain, nausea, vomiting, bleeding and laryngospasm .

Laryngospasm is a dangerous complication of tonsillectomy that occurs following tracheal extubation It is characterized by a strong, involuntary contraction of the laryngeal muscles, it's frequency in children is higher than adults due to their narrow upper airways that can be blocked following edema and inflammation The incidence of laryngospasm is 17 per 1000 children younger than nine years old, which increases to 96 per 1000 children with upper respiratory tract infections There are several ways to prevent this complication, including complete haemostasis during surgery, gentle suctioning of the oropharynx before extubation and the use of drugs as intravenous or topical lidocaine, propofol and etc .

Postoperative pain control after the tonsillectomy has a very important role in recovery time, hospitalization duration, bleeding, nausea and vomiting.

Lidocaine is an antiarrhythmic drug and its main mechanism of action is blocking voltage-gated Na+ channels that inhibit the activity of the upper laryngeal nerve and reduces the long-term blockage of the glottis .

Magnesium sulphate has a calcium antagonist property, which provides muscle relaxation and increases flaccidity. It also has an antagonistic action on sodium channels and N-methyl-D-aspartate receptors and reduces the release of substance P, which decreases the airway reactivity and stress responses .

Therefore we decided to compare the effect of intravenous injection of magnesium sulfate and lidocaine on the prevention of laryngospasm occurrence, and analgesic requirement in tonsillectomy the goal of the study Comparing the effectiveness of magnesium sulfate and lidocaine in prevention of post tonsillectomy complication .

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common surgeries in children which is associated with many morbidities such as postoperative pain, nausea, vomiting, bleeding and laryngospasm .

Laryngospasm is a dangerous complication of tonsillectomy that occurs following tracheal extubation It is characterized by a strong, involuntary contraction of the laryngeal muscles, it's frequency in children is higher than adults due to their narrow upper airways that can be blocked following edema and inflammation The incidence of laryngospasm is 17 per 1000 children younger than nine years old, which increases to 96 per 1000 children with upper respiratory tract infections There are several ways to prevent this complication, including complete haemostasis during surgery, gentle suctioning of the oropharynx before extubation and the use of drugs as intravenous or topical lidocaine, propofol and etc .

Postoperative pain control after the tonsillectomy has a very important role in recovery time, hospitalization duration, bleeding, nausea and vomiting.

Lidocaine is an antiarrhythmic drug and its main mechanism of action is blocking voltage-gated Na+ channels that inhibit the activity of the upper laryngeal nerve and reduces the long-term blockage of the glottis .

Magnesium sulphate has a calcium antagonist property, which provides muscle relaxation and increases flaccidity. It also has an antagonistic action on sodium channels and N-methyl-D-aspartate receptors and reduces the release of substance P, which decreases the airway reactivity and stress responses .

Therefore we decided to compare the effect of intravenous injection of magnesium sulfate and lidocaine on the prevention of laryngospasm occurrence, and analgesic requirement in tonsillectomy

ELIGIBILITY:
Inclusion Criteria:

* -ASA physical status I-II.
* Both sexes.
* Age: children 3-14years old.
* patients subjected for tonsillectomy or adeno-tonsillectomy surgery with parental consent for participation in the study.

Exclusion Criteria:

* - patients who refused to participate in this study.
* History of allergic response to magnesium sulfate and liodcaine .
* the Prescence of cardiovascular, respiratory and kidney diseases.
* A recent history of upper respiratory tract infection and febrile illness.
* History of mythenia gravis.
* patients subjected for adeno-tonsillectomy with myringotomy

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of laryngospasm in three groups. | 24 hours
  Common signs of laryngospasm include inspiratory stridor which may progress to complete obstruction, increased respiratory effort, tracheal tug, paradoxical respiratory effort, oxygen desaturation with or without bradycardia, or airway obstruction which does not respond to a Guedel airway. When these occur, either alone or in combination, laryngospasm is considered

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stalfors J, Ericsson E, Hemlin C, Hultcrantz E, Mansson I, Roos K, Hessen Soderman AC. Tonsil surgery efficiently relieves symptoms: analysis of 54 696 patients in the National Tonsil Surgery Register in Sweden. Acta Otolaryngol. 2012 May;132(5):533-9. doi: 10.3109/00016489.2011.644252. Epub 2012 Jan 11. PMID 22235871